CLINICAL TRIAL: NCT04426578
Title: Randomised Controlled Trial of pErhexiline on regreSsion Of Left Ventricular hypErtrophy (LVH) in Patients With Symptomatic Hypertrophic CardioMyopathy (RESOLVE-HCM)
Brief Title: Role of Perhexiline in Hypertrophic Cardiomyopathy
Acronym: RESOLVE-HCM
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Flinders University (Other)
Responsible Party: Principal Investigator, Joseph Selvanayagam, Professor, Flinders University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: HCM2020-01
Record Dates: First submitted 2020-05-14; First posted 2020-06-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Hypertrophic Cardiomyopathy
Keywords: Heart function and structure; Hypertrophy; Heart Failure; Medication; Imaging
MeSH Terms: conditions — Cardiomyopathy, Hypertrophic; Hypertrophy; Heart Failure | interventions — Perhexiline

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Perhexiline (Experimental)
  Interventions: Drug: Perhexiline
- Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: Perhexiline — All eligible and consented patients will be randomised to initiation of perhexiline 100mg once daily or identical placebo. After 4 days of treatment, a blood sample will be collected to determine plasma perhexiline concentrations: timing of the sample need not be "trough" in view of the long-acting nature of perhexiline. Depending on the blood results, patients might require as little as 50mg/week (slow metabolisers) or as much as 600mg/day (ultra-rapid metabolisers). The initial sample will be utilized primarily to detect presence of hydroxylated metabolite: patients in whom perhexiline is detected in the absence of metabolite will be designated "slow metabolisers" and will have their dosage reduced to 50 mg/week in the first instance. Repeat assay at 30 days will be utilized for individual finer dose titration based on dose adjustment table. Paired dosage adjustment in placebo-treated patients will be performed to avoid unblinding.
  Compliance will be assessed by capsule count.
  Other Names: Pexsig
  Arms: Perhexiline
Other: Placebo — All eligible and consented patients will be randomised to initiation of perhexiline 100mg once daily or identical placebo. After 4 days of treatment, a blood sample will be collected to determine plasma perhexiline concentrations: timing of the sample need not be "trough" in view of the long-acting nature of perhexiline. Depending on the blood results, patients might require as little as 50mg/week (slow metabolisers) or as much as 600mg/day (ultra-rapid metabolisers). The initial sample will be utilized primarily to detect presence of hydroxylated metabolite: patients in whom perhexiline is detected in the absence of metabolite will be designated "slow metabolisers" and will have their dosage reduced to 50 mg/week in the first instance. Repeat assay at 30 days will be utilized for individual finer dose titration based on dose adjustment table. Paired dosage adjustment in placebo-treated patients will be performed to avoid unblinding.
  Compliance will be assessed by capsule count.
  Arms: Placebo

SUMMARY:
Hypertrophic Cardiomyopathy (HCM) is the most common inherited heart muscle condition affecting up to 1 in 200 of the general population. It results from mutations in genes encoding components of the contractile apparatus in the heart muscle cell (myocyte). These mutations result in increased energy cost of force production for the myocyte which then cumulatively causes a myocardial energy deficit. This myocardial energy deficit is then thought to lead to cardiac hypertrophy ('left ventricular hypertrophy' or LVH) in HCM.

LVH leads to impairments in heart muscle function, heart muscle oxygenation and microvascular blood flow and is the chief driver of patient symptoms in HCM. These symptoms consist of chest pain, shortness of breath, dizziness, fainting episodes or palpitations. Occasionally, the disease may cause sudden cardiac death (SCD). HCM is the most common cause of SCD in young people including competitive athletes. In addition, HCM has been found to result in significant global deterioration in health-related quality of life.

Treatment of HCM has focused on relief of symptoms by drugs such as ß-blockers which slow the heart rate and improve heart function. However, symptom relief is often incomplete and there is no evidence on the benefit of ß-blockers or related medications to reverse LVH. Perhexiline, a potent carnitine palmitoyl transferase-1 (CPT-1) inhibitor shifts myocardial metabolism to more efficient glucose utilisation and rectifies impaired myocardial energetics. It is currently used to treat angina in patients with coronary artery disease. There is some preliminary evidence that Perhexiline may aid in the improvement of symptoms in patients with HCM. However, the effect of any form of therapy on potential regression of LVH in HCM remains unexplored.

In this randomised double-blind placebo-controlled trial, the investigators will use state of the art cardiac imaging, principally advanced echocardiography and Cardiovascular Magnetic Resonance (CMR) to study the effects of perhexiline on LVH, cardiac function, and oxygenation in symptomatic patients with HCM. The investigators hypothesize that perhexiline will favourably reduce LVH and improve myocardial oxygenation by improving myocardial energetics, and that these putative morphological and functional changes can be accurately measured utilizing echocardiography and CMR. If this pilot study supports the hypothesis, then it will pave the way for a major randomised controlled trial to definitely determine the role of Perhexiline in HCM.

ELIGIBILITY:
Inclusion Criteria:

1. Left Ventricular Ejection Fraction (LVEF) =/> 55% by echocardiography or CMR during the screening period or within 6 months prior to study entry
2. Current / prior symptom(s) of HCM (New York Heart Association [NYHA] functional class II or class III, Canadian Cardiovascular Society [CCS] grade II or grade III) and requiring treatment with ß-blockers and /or non-dihydropyridine calcium antagonists and / or disopyramide for at least 30 days prior to study entry
3. Structural heart disease as evidenced by interventricular septal thickness of (= 15 mm) on echocardiography or CMR in the absence of abnormal loading conditions
4. Elevated N terminal pro-brain natriuretic peptide (NT-proBNP), >125 pg/ml

Exclusion Criteria:

1. Any prior echocardiographic or CMR measurement of LVEF <55%
2. Current acute decompensated heart failure requiring hospitalisation and / or augmented medical therapy
3. Cardiac surgery or catheter-based septal reduction therapy planned or having occurred within the past 1 year
4. Patients with a non-CMR conditional pacemaker / implantable cardioverter-defibrillator device
5. History of a known chronic liver disease, peripheral neuropathy, recurrent hypoglycemia
6. Serum bilirubin, alanine aminotransferase, aspartate aminotransferase, alkaline phosphatase, or lactate dehydrogenase > 2.0 times upper limit of normal
7. Previous adverse reaction to perhexiline at therapeutic plasma levels of the drug
8. Concomitant use of amiodarone, ranolazine or trimetazidine
9. Life-threatening or uncontrolled dysrhythmia
10. Contraindications to CMR, gadolinium, adenosine

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-12-01 (Actual); Primary Completion 2022-08-01 (Estimated); Study Completion 2022-08-01 (Estimated)

PRIMARY OUTCOMES:
Change in Left Ventricular Hypertrophy (LVH) | 12 months post baseline
  Change in LVH (septal thickness) in symptomatic at 12 months following perhexiline therapy in HCM patients assessed by CMR

SECONDARY OUTCOMES:
Change in Left Ventricular (LV) mass | 12 months post baseline
  Change in left ventricular mass in symptomatic at 12 months following perhexiline therapy in HCM patients assessed by CMR
Change in oxygen-sensitive Cardiac Magnetic Resonance | 12 months post baseline
  Change in oxygen-sensitive CMR in symptomatic at 12 months following perhexiline therapy in HCM patients
Change in left ventricular diastolic function | 12 months post baseline
  Change in left ventricular diastolic function at 12 months following perhexiline therapy in HCM patients assessed by echocardiography
New York Heart Association (NYHA) functional classification | 12 months post baseline
  Change in NYHA classification of Class I, II, III and IV at 12 months following perhexiline therapy in HCM patients
Canadian Cardiovascular Society (CCS) functional class | 12 months post baseline
  Change in CCS functional classification of Grade I, II, III and IV at 12 months following perhexiline therapy in HCM patients
Quality of life assessment | 12 months post baseline
  Change in physical activity domain score of Short Form 36 Health Survey Questionnaire (SF36) at 12 months following perhexiline therapy in HCM patients
Major adverse event on heart failure related hospitalisations | Monitored over the 12 months period
  HCM patients admitted with heart failure during the study period
Major adverse event on arrhythmic events | Monitored over the 12 months period
  HCM patients admitted with arrhythmic events during the study period
Major adverse event on abnormal liver function test | Liver function tests at baseline, 1 month, 6 months and 12 months
  HCM patients with abnormal liver function tests during the study period
Major adverse event on sudden cardiac death | Monitored over the 12 months period
  HCM patients with sudden cardiac death during the study period

CONTACTS AND LOCATIONS:
Overall Officials: Joseph Selvanayagam, Study Chair — Flinders Medical Centre; Rajiv Ananthakrishna, Principal Investigator — Flinders Medical Centre
Locations (1):
- Flinders Medical Centre, Adelaide, South Australia, Australia

IPD SHARING:
Plan to Share IPD: No